CLINICAL TRIAL: NCT00612937
Title: Respiratory Distress of the Newborn and Its Relationship to Group B Streptococcal Colonization
Brief Title: Streptococcal Infection and Respiratory Distress in Newborns
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999908069; 08-CH-N069
Record Dates: First submitted 2008-02-10; First posted 2008-02-12 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2015-06-19

CONDITIONS: Group B Streptococci; Respiratory Distress in Newborn
Keywords: Group B Streptococci; Respiratory Disease; Beta Lactam; Newborn; Respiratory Distress
MeSH Terms: conditions — Respiration Disorders; Dyspnea

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study will evaluate whether babies are more at risk of developing breathing problems if their mothers carry group B streptococci (GBS) in vagina/rectum, and whether the breathing problem is due to phospholipids released by the GBS. About one in five pregnant women carry GBS in their vagina/rectum. Mothers who carry these bacteria are given antibiotics during labor to prevent infection in the baby. However, recently it has been suspected that even without blood stream infection, the chemicals released by GBS, called phospholipids, might lead to breathing problems.

Women at 32 or more weeks of pregnancy who deliver at Ben Taub Hospital and St. Luke s Episcopal Hospital in Houston, Texas, and Alta Bates Summit Medical Center in Oakland, California, may be eligible for this study.

Mothers undergo the following procedures:

* Vaginal/rectal GBS culture. A sample is collected from the lower vagina and rectum using a cotton swab upon admission to labor and delivery.
* Blood collection to test for phospholipids. A blood sample is obtained from the mothers at the time of routine blood drawing during labor, and a blood sample is obtained from the umbilical cord (after delivery).
* Collection of health information from the medical record.

Newborns undergo the following procedures:

* GBS culture. Samples are collected from cotton swabs of the ears, navel, anus and throat to test for GBS bacteria.
* A small amount of blood from newborns is obtained for phospholipids test when the newborns have blood drawn for other tests.
* Collection of health information from the medical record.

DETAILED DESCRIPTION:
Phospholipids from the group B streptococcal (GBS) cell wall cause pulmonary hypertension in experimental animals. We hypothesize that newborns colonized with GBS receive bacterial phospholipids leading to pulmonary hypertension and respiratory distress. When exposed to penicillin (beta-lactam), Streptococcus mutans releases phospholipids immediately. An analysis of 1610 colonized newborns from the NICHD GBS study conducted in six academic centers from 1995 to 1999 showed that 8.8% of GBS colonized newborns greater than or equal to 32 weeks gestation had signs of respiratory distress as compared to 1-3% observed in general newborn populations, and that beta-lactam use during labor was associated with 2.62 fold increase in respiratory distress in the colonized newborns. These findings support the association of neonatal respiratory distress with GBS colonization and with penicillin use during labor. These data however require confirmation.

We now plan to conduct a prospective study to relate the levels of serum bacterial phospholipids to the occurrence of respiratory distress in newborns of mother colonized GBS. This study will also evaluate the effect of beta-lactam use during labor on the release of phospholipids and therefore the occurrence of respiratory distress in newborns of mothers colonized with GBS. The study will be conducted at the Baylor College of Medicine and Oakland Children s Hospital and Research Center. Serum phospholipid levels will be measured in newborns with respiratory distress, newborns of mothers colonized by GBS, treated or untreated with beta-lactam during labor.

ELIGIBILITY:
* INCLUSION CRITERIA:

All women who are admitted to labor and delivery room at greater than or equal to 32 weeks gestation will be approached for obtaining consent to participate in this study.

EXCLUSION CRITERIA:

Newborns with severe or fatal congenital anomaly such as gastroschisis, congenital diaphragmatic hernia, tracheoesophageal fistula, transition of the great arteries, coarctation of aorta, myelomeningocele, and omphalocele will be excluded from the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13180 (Actual)
Dates: Start 2008-02-04; Study Completion 2015-06-19

CONTACTS AND LOCATIONS:
Overall Officials: Forbes D Porter, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (2):
- United States (2):
  - Oakland Children's Hospital and Research Center, Oakland, California
  - Baylor College of Medicine, Houston, Texas

REFERENCES:
- [Background] McCracken GH Jr. Group B streptococci: the new challenge in neonatal infections. J Pediatr. 1973 Apr;82(4):703-6. doi: 10.1016/s0022-3476(73)80603-1. No abstract available. PMID 4572746
- [Background] Katzenstein AL, Davis C, Braude A. Pulmonary changes in neonatal sepsis to group B beta-hemolytic Streptococcus: relation of hyaline membrane disease. J Infect Dis. 1976 Apr;133(4):430-5. doi: 10.1093/infdis/133.4.430. PMID 57196
- [Background] Weisman LE, Stoll BJ, Cruess DF, Hall RT, Merenstein GB, Hemming VG, Fischer GW. Early-onset group B streptococcal sepsis: a current assessment. J Pediatr. 1992 Sep;121(3):428-33. doi: 10.1016/s0022-3476(05)81801-3. PMID 1517922